CLINICAL TRIAL: NCT05476341
Title: A Randomized, Double-blind, Single Dose, Parallel Comparison of Bevacizumab Injection and Avastin ® Phase I Clinical Study on the Similarity of Pharmacokinetics and Safety of Traditional Chinese Medicine in Healthy Male Volunteers
Brief Title: A Phase I Clinical Trial of Bevacizumab Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDTQ-2017-BFZDK
Record Dates: First submitted 2022-07-18; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Rectal Cancer; Lung Cancer; Ovarian Cancer; Cervical Cancer; Glioblastoma
MeSH Terms: conditions — Rectal Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Glioblastoma | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab injection (Experimental): On the first day, bevacizumab injection was given, 3mg/kg each time, diluted to 100ml of 0.9% sodium chloride injection, mixed evenly, and then intravenous infusion for 90 minutes (±15 minutes).
  Interventions: Drug: Bevacizumab injection
- Bevacizumab injection（Avastin） (Active Comparator): On the first day, Avastin injection was given, 3mg/kg of which was diluted to 100ml of 0.9% sodium chloride injection. After mixing evenly, it was infused intravenously for 90 minutes (±15 minutes).
  Interventions: Drug: Bevacizumab injection（Avastin）

INTERVENTIONS:
Drug: Bevacizumab injection — Recombinant humanized monoclonal antibody injection against human vascular endothelial growth factor
  Arms: Bevacizumab injection
Drug: Bevacizumab injection（Avastin） — Recombinant humanized monoclonal antibody injection against human vascular endothelial growth factor
  Arms: Bevacizumab injection（Avastin）

SUMMARY:
Recombinant humanized monoclonal antibody injection against human vascular endothelial growth factor (bevacizumab) is Avastin produced by Zhengda Tianqing Pharmaceutical Group Co., Ltd Biological similar drugs. Its mechanism is to prevent VEGF from binding to its natural receptor VEGFR, inhibit the proliferation and activation of vascular endothelial cells, and play an anti angiogenesis and anti-tumor role by binding with VEGF. A randomized, double-blind, single dose, parallel comparison of bevacizumab injection and Avastin is planned The phase I clinical study on the similarity of pharmacokinetics and safety of traditional Chinese medicine in healthy male volunteers aims to compare bevacizumab injection with Avastin The similarity of pharmacokinetics, tolerance, safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* 1 Fully understand the purpose of the test, and basically understand the pharmacological effects and possible adverse reactions of the research drugs; Voluntarily sign written informed consent in accordance with the spirit of the Helsinki declaration.
* 2 Healthy male subjects aged ≥ 18 and ≤ 65.
* 3 Weight ≥ 50 kg and ≤ 80 kg, body mass index (BMI) ≥ 18 and ≤ 28kg/m2.
* 4 Each system examination index is within the normal range, or the examination result is abnormal, but it is judged by the researcher to be of no clinical significance.
* 5 The subjects agreed to use reliable contraceptives for themselves and their partners during the study period and within 6 months after the infusion of the study drug(such as abstinence, sterilization, contraceptive pills, injection of contraceptive medroxyprogesterone or subcutaneous implantation contraception, etc).

Exclusion Criteria:

* 1 Have a history of hypertension or abnormal blood pressure during screening / baseline measurement(Repeated measurements on the same day confirmed that systolic blood pressure [SBP] > 140 mmHg and / or diastolic blood pressure [DBP] > 90 mmHg).
* 2 Clinically significant proteinuria (routine urine examination, urine protein 2+ and above) or history of proteinuria assessed by the investigator.
* 3 Have received any antibody or protein therapy targeting VEGF or VEGF receptor in the past 1 year.
* 4 Used any biological products or vaccinated with live virus vaccine within 3 months before the infusion of the study drug, or used any monoclonal antibody within 12 months.
* 5 Have hereditary bleeding tendency or coagulation dysfunction, or have a history of thrombosis or bleeding.
* 6 Have a history of gastrointestinal perforation or fistula.
* 7 Unhealed wound ulcer or fracture, or major surgery within the first 2 months of randomization, or major surgery expected during the study period or within 2 months after the end of the study.
* 8 Use prescription or over-the-counter drugs or nutritional health products, and the use time is within 5 half lives of the drugs or nutritional health products or within 2 weeks before the use of the study drugs (the time limit is whichever is longer).Herbal health products should be stopped 28 days before using the study drug.
* 9 Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody or syphilis antibody are tested positive.
* 10 Known allergy to bevacizumab or any of its excipients.
* 11 People with known history of allergic diseases or allergic constitution.
* 12 There was a history of blood donation 3 months before the infusion of the study drug.
* 13 Have been treated with any other research drugs or participated in another intervention clinical trial within 2 months before screening.
* 14 Have a history of alcohol or drug abuse within 12 months before screening; The subjects were unable to quit drinking within 72 hours before administration and throughout the trial.
* 15 Have a history of mental illness.
* 16 Subjects whose spouses plan to conceive.
* 17 Unable to follow the protocol requirements to complete the study during the study.
* 18 Other researchers think it is not suitable to be included in the group

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Plasma concentration-area under time curve（AUC0-t） | Within 30 minutes before administration to 1680 hours (day 71)
  Area under the blood concentration time curve from 0 hour to the collection time t of the last measurable concentration

SECONDARY OUTCOMES:
Plasma concentration-area under time curve（AUC0-∞） | Within 30 minutes before administration to 1680 hours (day 71)
  Area under the blood concentration time curve from 0 hour to inf (infinity)
Peak concentration (Cmax) | Within 30 minutes before administration to 1680 hours (day 71)
  Maximum plasma concentration observed after administration
Incidence of adverse events | Within 30 minutes before administration to 1680 hours (day 71)
  Incidence of adverse events assessed by CTCAE v4.0
Number of adverse events related to the study drug | Within 30 minutes before administration to 1680 hours (day 71)
  Number of adverse events evaluated by CTCAE v4.0
Incidence of adverse events related to the study drug | Within 30 minutes before administration to 1680 hours (day 71)
  Incidence of study drug-related adverse events assessed by CTCAE v4.0
ADA positive rate | Within 30 minutes before administration to 1680 hours (day 71)
  When anti drug antibody (ADA) is positive, neutralizing antibody (NAB) test is performed

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China